CLINICAL TRIAL: NCT00355953
Title: Vascular and Skeletal Protective Effects of Genistein in Postmenopausal Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Messina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002067398
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Menopause; Osteopenia
Keywords: Post-Menopausal Women; Osteoporosis; Phytoestrogen; Genistein
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Genistein

INTERVENTIONS:
Drug: Genistein

SUMMARY:
The present research program is proposed deepening some pharmacological effects of the genistein therapy in order to individualize alternative treatments to the conventional hormonal replacement therapy useful to reduce the cardiovascular morbidity and mortality and the osteoporotic consequences in postmenopausal women.

DETAILED DESCRIPTION:
Genistein is a phytoestrogen of the isoflavone family which has been shown to have beneficial effects on endothelial function and bone metabolism. On the basis of the so far obtained results, aim of our research was to investigate for a two years period the effects of genistein on cardiovascular risk factors, endothelial function and oxidative stress markers, bone metabolism and finally clarify pathophysiology mechanisms (by dosage of cytokines and endothelial markers) by which this molecule could interfere on atherosclerosis and bone mass loss progression.

Particularly, and in extreme synthesis the following parameters have been studied during the treatment:

1. inflammation markers as fibrinogen
2. lipid profile - total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, lipoprotein(a)-
3. endothelial function markers as VCAM-1 and ICAM-1
4. oxidative stress by the evaluation of the F(2)-isoprostane
5. cytokines as IL-6, OPG, RANK and RANKL
6. bone mineral density, by DEXA, at lumbar spine and femoral neck
7. Bone turnover markers as B-ALP, PYR, D-PYR
8. PAP-test, transvaginal uterine ecography and mammography.

ELIGIBILITY:
Inclusion Criteria:

* At least one year of menopause
* No use of hormone replacement therapy
* Bone mineral density T-score at the femoral neck minor than one S.D.

Exclusion Criteria:

* Concomitant disease
* Smoke habit

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-01; Study Completion 2005-06

PRIMARY OUTCOMES:
Efficacy:
bone resorption/formation
bone mineral density
cardiovascular risk factors
Safety:
endometrial thickness

SECONDARY OUTCOMES:
Efficacy:
hot flushes reduction
Safety:
mammography
vaginal cells maturation value

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Squadrito, MD, Study Director — University of Messina

REFERENCES:
- [Derived] Marini H, Minutoli L, Polito F, Bitto A, Altavilla D, Atteritano M, Gaudio A, Mazzaferro S, Frisina A, Frisina N, Lubrano C, Bonaiuto M, D'Anna R, Cannata ML, Corrado F, Adamo EB, Wilson S, Squadrito F. Effects of the phytoestrogen genistein on bone metabolism in osteopenic postmenopausal women: a randomized trial. Ann Intern Med. 2007 Jun 19;146(12):839-47. doi: 10.7326/0003-4819-146-12-200706190-00005. PMID 17577003